CLINICAL TRIAL: NCT07253792
Title: The Effect of Cancer Screening Training Provided to Academics at a Foundation University on Cancer Screening Knowledge Levels and Family Health Center Utilization Rates
Brief Title: Cancer Screening Training for Academics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Responsible Party: Principal Investigator, Naciye Esra Koyuncu, Researcher Assistant, KTO Karatay University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 14.04.2025-E.107676
Record Dates: First submitted 2025-08-01; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Cancer
Keywords: Health Education; knowledge; Primary Health Care; Health Professional; Nursing
MeSH Terms: conditions — Neoplasms; Health Education

STUDY DESIGN:
Intervention Model Description: Pre-test data, including the Personal Information Form and the Cancer Screening Information Scale, were collected from participants in the intervention group before the training began. The pre-test took approximately 5-10 minutes to complete. Subsequently, this group received training on cancer screening and Family Health Centre use once a week for a total of four weeks. Following the completion of the training, a post-test was administered at the end of the fourth week.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Pre-test data, including the Personal Information Form and the Cancer Screening Information Scale, were collected from participants in the intervention group before the training began. The pre-test took approximately 5-10 minutes to complete. Subsequently, this group received training on cancer screening and Family Health Centre use once a week for a total of four weeks. Following the completion of the training, a post-test was administered at the end of the fourth week.
  Interventions: Behavioral: Cancer training
- control (No Intervention): No training was provided to participants in the control group. Participants in this group were only asked to complete a Personal Information Form at the beginning of the study, and final test data was collected at the end of the four weeks.

INTERVENTIONS:
Behavioral: Cancer training — Pre-test data, including the Personal Information Form and the Cancer Screening Information Scale, were collected from participants in the intervention group before the training began. The pre-test took approximately 5-10 minutes to complete. Subsequently, this group received training on cancer screening and Family Health Centre use once a week for a total of four weeks. Following the completion of the training, a post-test was administered at the end of the fourth week.
  Arms: Intervention

SUMMARY:
Purpose: The purpose of this research is to examine the effect of cancer screening education on individuals' knowledge levels regarding cancer screening and their rates of utilization of primary health care services.

Method: The research was conducted using a parallel group pretest-posttest experimental design. The study, conducted at a foundation university between April and May 2025, included 71 academics selected using simple random sampling. The intervention group received structured cancer screening education for four weeks. Data will be collected using a Personal Information Form and the Cancer Screening Knowledge Scale (CSKS), and will be analyzed using appropriate statistical methods.

ELIGIBILITY:
Inclusion Criteria:

* Be employed full-time at the university,
* Be able to read and understand Turkish,
* Not have received any cancer screening training in the last 6 months

Exclusion Criteria:

* Those who did not participate in the training or participated incompletely,
* Those with incomplete information in the pre-test or post-test data,
* Those who have been diagnosed with cancer and are undergoing treatment

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Family health centre utilisation rate | From baseline to 1 month post-training
  Family health centre utilisation rate: The proportion of participants who report using services provided by a family health centre within a specified time frame. This includes visits for preventive care, screening, diagnosis, treatment, or follow-up services, as defined by the study protocol.
Cancer knowledge level | From baseline to 1 month post-training
  Cancer knowledge level: The score obtained from the Cancer Screening Knowledge Scale (CSKS), which measures participants' knowledge about cancer screening methods, recommended screening intervals, and target populations. Higher scores indicate a greater level of knowledge, as defined by the study protocol.

CONTACTS AND LOCATIONS:
Locations (1):
- KTO Karatay University, Konya, Akabe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
"Individual participant data will not be shared due to privacy concerns and institutional ethical restrictions. The dataset includes identifiable information that cannot be fully anonymized.

REFERENCES:
- [Background] Dagar, M., Upadhyay, P., & Kumar, P. (2025). Assessing Cancer Awareness and Knowledge Among Healthcare Professionals in a Tertiary Care Teaching Hospital, Bareilly. SRMS JOURNAL OF MEDICAL SCIENCE, 10(Suppl1), S13-S19. https://doi.org/10.21761/JMS.V10ISUPPL.04